CLINICAL TRIAL: NCT07240857
Title: A Clinical Study Evaluating the Safety and Efficacy of Local Injection of ACT#001 Chimeric Antigen Receptor T Cells in the Treatment of Castration-Resistant Prostate Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Orig Stone Biotech(Zhejiang) Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACT#001
Record Dates: First submitted 2025-08-23; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Castration-Resistant Prostate Cancer (CRPC)
Keywords: CAR-T; CRPC
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid titration dose exploration phase (Experimental): It is 18×10⁶ CAR-T cells, and it is planned to include 1 participant,If the participant experiences no dose-limiting toxicity (DLT) or grade 2 adverse reactions, the dose will be escalated to the 5×10⁷ CAR-T cells group for the "3+3" dose escalation; if the patient develops DLT or grade 2 adverse reactions, 2 additional participants will be enrolled, and the study will switch to the traditional "3+3" design for dose exploration.
  Interventions: Biological: Intraprostatic or localized lesion injection of ACT#001-PSMA CAR-T cells under transrectal ultrasound (TRUS) guidance
- "3+3" dose escalation phase (Experimental): Dose escalation will be conducted sequentially in two dose groups: 5×10⁷ CAR-T cells and 1×10⁸ CAR-T cells. In view of the particularity of cell preparations, the actual administration dose in each dose group is allowed to have a fluctuation of ±30%.
  Each dose group will first enroll 3 participants. Within the same dose group, the interval between cell infusions for the first 2 participants should not be less than 14 days. During dose escalation, the interval between the infusion time of the last participant in each dose level and that of the first participant in the next dose level should be at least 28 days.If no dose-limiting toxicity (DLT) is observed in all participants within the same dose group, the dose will be escalated to the next level. If 1 case of DLT occurs, 3 additional participants will be enrolled in this dose group (with a total of 6 participants enrolled). If no new DLT occurs, the dose will be escalated to the next level.
  Interventions: Biological: Intraprostatic or localized lesion injection of ACT#001-PSMA CAR-T cells under transrectal ultrasound (TRUS) guidance

INTERVENTIONS:
Biological: Intraprostatic or localized lesion injection of ACT#001-PSMA CAR-T cells under transrectal ultrasound (TRUS) guidance — Prior to CAR-T cell infusion, subjects will receive lymphodepleting chemotherapy based on fludarabine and cyclophosphamide.
  Surgical method :
  1)The patient is taken to the operating room, and the anesthesia method is intravenous anesthesia or local anesthesia. A digital rectal examination is performed, and the anus is dilated to accommodate three fingers. The genitals and perineum are prepared and covered in a sterile manner. An ultrasound probe is inserted into the rectum; (2) Under ultrasound guidance, CAR-T cells are injected into the prostate or localized lesions via the rectum or perineum; (3) Then, the TRUS probe is removed from the patient's rectum.

SUMMARY:
An exploratory clinical study evaluating the safety and efficacy of ACT#001 chimeric antigen receptor T-cell (CAR-T cell) local injection in the treatment of castration-resistant prostate cancer.

DETAILED DESCRIPTION:
Chimeric Antigen Receptor (CAR) T cells are genetically engineered T cells that can express the introduced CAR gene, which contains signaling molecules such as antigen recognition fragments, T cell receptor activation molecules, and co-stimulatory signals. Currently, in the field of hematological tumors, CD19-targeted CAR-T cells have been clinically proven to effectively treat B-cell malignancies. The US FDA has approved their use for treating relapsed or refractory CD19-positive B-cell malignancies, with favorable therapeutic effects. However, significant challenges remain before CAR-T therapy can be widely applied to solid tumor treatment. For example, the non-specific targeting of CAR-T cells to normal/non-malignant tissues ("on-target, off-tumor toxicity") can be fatal. In fact, off-tumor toxicity to the lungs, cerebral gray matter, and cardiac muscle has resulted in multiple deaths.

Prostate-specific membrane antigen (PSMA) is a surface antigen highly expressed in prostate cancer. Over 98% of lymph node metastases and almost all bone metastases in patients with castration-resistant prostate cancer (CRPC) highly express PSMA, making it an ideal target for prostate cancer treatment. We have developed a thermally activated and regulated FB-PSMA CAR-T cell targeting the prostate cancer antigen PSMA. In vitro, heating at 43°C can activate CAR expression without impairing cell function. After injection into the tumor site, PSMA-expressing prostate cancer cells can activate FB-PSMA CAR-T cells and, through a feedback mechanism, increase the expression level of CAR molecules, thereby enhancing the tumor-killing effect. Once tumor elimination is completed, CAR molecules will gradually degrade to provide a higher level of safety. In a mouse model of prostate cancer xenografts, FB-PSMA CAR-T cells have demonstrated significant anti-tumor effects and good safety.

Based on the above background, we plan to conduct this clinical trial, aiming to explore a new immunotherapeutic approach that can effectively control prostate cancer while maximizing the preservation of urogenital function and the control of oligometastases, thereby addressing the unmet needs in the current treatment of local prostate cancer. We hope that through this study, we can provide a safer and more effective treatment option for prostate cancer patients, while opening up new possibilities for future cancer treatment. This study is designed to evaluate the safety and efficacy of local injection of ACT#001 chimeric antigen receptor T cells (ACT#001-PSMA CAR-T) in the treatment of castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria

1. understanding of this study and voluntarily signs the informed consent form;
2. Aged ≥ 18 years;
3. Expected survival time of at least 3 months;
4. non-metastatic CRPC (nmCRPC) (local recurrence) or metastatic CRPC (mCRPC)；
5. continue GnRH analog therapy；
6. at least one evaluable lesion per RECIST 1.1;
7. Has received at least one type of novel endocrine therapy；
8. PSMA positive expression rate > 10%;
9. Eastern Cooperative Oncology Group (ECOG) 0-1;
10. Well organ function
11. Left Ventricular Ejection Fraction (LVEF) > 50%;
12. Oxygen saturation > 92% without oxygen supplementation;
13. agree to use effective contraceptive measures

Exclusion Criteria

1. Presence of brain metastasis;
2. Organ transplantation or pending organ transplantation;
3. Uncontrolled large-volume serous cavity effusions；
4. A history of autoimmune diseases；
5. A history of receiving other cell therapies or genetically modified cell therapies (e.g., TCR-T therapy, CAR-T therapy);
6. A history of receiving any PSMA-targeted therapy;
7. Requirement for steroid therapy (except for physiological replacement therapy);
8. A history of receiving immunotherapies;
9. A history of clinically significant central nervous system (CNS) diseases (either past or present at screening);

(12) A history of other untreated malignant tumors; (13) Participants with severe cardiovascular diseases; (14) Active infectious diseases; (15) Active hepatitis B or hepatitis C virus infection; (16) Active Epstein-Barr virus (EBV) or cytomegalovirus (CMV) infection (17) Intolerance or allergy to cyclophosphamide or fludarabine chemotherapeutic drugs; (18) No accessible injection sites; (19) Assessment by the investigator that the participant is unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  adverse events occurring within 28 days after the first infusion that are related to the study drug (definitely related, probably related, possibly related).

SECONDARY OUTCOMES:
PSA50 response rate | 6 months
  The proportion of participants with a reduction of ≥50% in PSA from baseline to the lowest post-baseline PSA result, which needs to be confirmed by a second consecutive PSA assessment after at least 3 weeks.
DoPSA50（duration of PSA50 response） | 6 months
  The time from the date of first documented PSA50 response (subsequently confirmed) to the date of documented PSA progression per PCWG3 criteria or death from any cause in the absence of PSA progression.
DRRPSA50（durable PSA50 response rates） | 6 months
  The percentage of participants with a confirmed PSA50 response lasting at least 6 months, using the number of participants in the PSA evaluable set as the denominator.
TTPSAP50（time to PSA50 progression ) | 6 months
  The time from the date of the first documented PSA50 response (subsequently confirmed) to the date of documented PSA progression per PCWG3 criteria.
PSA90 response rate | 6 Months
  The proportion of participants with a reduction of ≥90% in PSA from baseline to the lowest post-baseline PSA result, which needs to be confirmed by a second consecutive PSA assessment after at least 3 weeks.
DoPSA90（duration of PSA90 response） | 6 months
  The time from the date of first documented PSA90 response (subsequently confirmed) to the date of documented PSA progression per PCWG3 criteria or death from any cause in the absence of PSA progression.
DRRPSA90（durable PSA90 response rates) | 6 months
  The percentage of participants with a confirmed PSA90 response lasting at least 6 months, using the number of participants in the PSA evaluable set as the denominator.
TTPSAP90（time to PSA90 progression) | 6 months
  The time from the date of the first documented PSA90 response (subsequently confirmed) to the date of documented PSA progression per PCWG3 criteria.
ORR | 6 MONTHS
  The proportion of patients achieving complete response (CR) or partial response (PR).
DOR（Duration of Response） | 6MONTHS
  The duration from the initial achievement of partial response (PR) or complete response (CR) to the occurrence of disease progression or death.
DCR（Disease Control Rate） | 6months
  The proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD).
TTR（Time to Response） | 6mohths
  The time from treatment initiation to the first achievement of partial response (PR) or complete response (CR).
OS（Overall Survival） | 6 months
  The time from treatment initiation to death from any cause.
rPFS（Radiographic Progression-Free Survival） | 6 months
  The time from treatment initiation to radiologically documented disease progression or death.
mFS | 6 months
  The time from treatment initiation to the development of distant metastasis or death.
In vivo persistence time of CAR-T cells | 6 months
  The time from the infusion of ACT#001-PSMA CAR-T cells to the point when ACT#001-PSMA CAR-T cells can no longer be detected in the body (with 2 consecutive negative test results), which is detected by methods such as QPCR and flow cytometry.

OTHER OUTCOMES:
The proportion of immune cell subsets in peripheral blood | 28 DAYS
  At five fixed timepoints-pre-lymphodepletion, post-lymphodepletion (pre-infusion), post-infusion (D0/D1), discharge (e.g., D7), and D28-as well as at the onset of CRS, to explore the proportion of immune cell subsets in peripheral blood
The proportion of subgroups of the intestinal microbiota | 28 DAYS
  At five fixed timepoints-pre-lymphodepletion, post-lymphodepletion (pre-infusion), post-infusion (D0/D1), discharge (e.g., D7), and D28-as well as at the onset of CRS to explore the the proportion of subgroups of the intestinal microbiota from stool samples
The correlation between therapeutic effect and PSA level | 6 months
  The correlation between therapeutic effect and PSA level
The correlation between therapeutic effect and percentage of histological PSMA expression | 6 months
  The correlation between therapeutic effect and percentage of histological PSMA expression
The correlation between therapeutic effect and HRR mutation status | 6 months
  The correlation between therapeutic effect and HRR mutation status
The correlation between therapeutic effect and dMMR/MSI-H status | 6 months
  The correlation between therapeutic effect and dMMR/MSI-H status
The correlation between therapeutic effect and prior treatment regimens | 6 months
  The correlation between therapeutic effect and prior treatment regimens
The correlation between therapeutic effect and disease classification (mCRPC vs. nmCRPC) | 6 months
  The correlation between therapeutic effect and disease classification (mCRPC vs. nmCRPC)